CLINICAL TRIAL: NCT01135654
Title: Alcohol SBIRT Implementation in an HMO: Non-Physician Providers Vs Physicians
Brief Title: Alcohol Drinking as a Vital Sign
Acronym: ADVISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CN-09JMert-03-H; R01AA018660 (NIH)
Record Dates: First submitted 2010-06-01; First posted 2010-06-03 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Unhealthy Drinking; Alcohol Dependence
Keywords: alcohol dependence; unhealthy drinking; SBIRT
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; Mass Screening; Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Non-Physician Provider (Experimental)
  Interventions: Other: Training & Tech Support for Delivery of Alcohol Screening, Brief Intervention, and Referral To Treatment
- Control (No Intervention)
- Primary Care Provider (Active Comparator): In clinics randomized to this arm, we will train (and provide technical assistance to) Primary Care providers to conduct Alcohol Screening, Brief Intervention, and Referral to Treatment.
  Interventions: Other: Training & Tech Support for Delivery of Alcohol Screening, Brief Intervention, and Referral To Treatment

INTERVENTIONS:
Other: Training & Tech Support for Delivery of Alcohol Screening, Brief Intervention, and Referral To Treatment — We provide training and technical support for providers to conduct Alcohol Screening, Brief Intervention, and Referral to Treatment. The training is based on the NIAAA clinician's guide to "Helping Patients Who Drink Too Much".
  Arms: Non-Physician Provider; Primary Care Provider

SUMMARY:
The purpose of this study is to determine whether Alcohol Screening, Brief Intervention, and Referral to Specialty Chemical Dependency Treatment (as appropriate) by Non-Physicians versus Primary Care Providers (versus control group) is more likely to be implemented and more effective at reducing unsafe drinking.

DETAILED DESCRIPTION:
This health services implementation study is a clustered, randomized trial. We propose to randomize primary care clinics to three arms-a control condition and two alternative modes of delivery of the NIAAA Clinician's Guide to Alcohol Screening, Brief Intervention, and Referral to Treatment (SBIRT) in primary care settings. In the Primary Care Physician or "PCP" arm, PCPs will be trained on the SBIRT protocols outlined in the NIAAA Clinicians' Guide and conduct brief intervention and referrals as needed. In the Non-Physician Provider or "NPP" arm, Medical Assistants will be trained to use the NIAAA screener and enter the results in the Electronic Medical Record, and NPPs (e.g., Behavioral Medicine Specialists, Clinical Nurses and Health Educators) will conduct brief intervention and referral activities. The SBIRT content, based on the NIAAA Guide, is the same in both the NPP and PCP arms; we compare delivery by the two types of providers and versus the control condition, in which providers and staff will not receive any training on SBIRT protocols. We examine implementation outcomes: rates of screening, brief intervention, follow-up screening and brief intervention, referral to Chemical Dependency treatment, and alcohol use disorders medication rates. We also include, as secondary analyses, an effectiveness study examining patient outcomes by study arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients: All patients aged 18+ who receive primary care visits in the Kaiser Permanente clinics in Northern California.

Exclusion Criteria:

* Patients younger than 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 639613 (Actual)
Dates: Start 2010-01; Primary Completion 2012-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients screened for alcohol | One year
  We define the Screening Rate as the proportion of patients who receive the NIAAA brief screener (available in the Electronic Medical Record) from among all unique patients who have visits to the clinics in the relevant study arm in the year following the training of providers.
Proportion receiving Brief Intervention among those who screen positive to screener. | One year.
  The proportion receiving Brief Intervention Rate is the proportion of patients who receive brief intervention from among all patients who have visits to the clinic in the one year period and screen positive on the NIAAA screener in the EMR.
Proportion of patients referred to treatment | one year
  The treatment referral rate will be defined as the proportion of patients who receive referrals to Chemical Dependency treatment from among those who receive alcohol dependence diagnoses or whose screener indicates possible alcohol dependence.

SECONDARY OUTCOMES:
Changes in quantity of alcohol consumption - average weekly consumption | one year
  We will examine changes in alcohol consumption measures (average weekly consumption at subsequent visits) for those who have return visits within the study observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Sterling, DrPH, MSW, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northern California, Oakland, California, United States

REFERENCES:
- [Derived] Mertens JR, Chi FW, Weisner CM, Satre DD, Ross TB, Allen S, Pating D, Campbell CI, Lu YW, Sterling SA. Physician versus non-physician delivery of alcohol screening, brief intervention and referral to treatment in adult primary care: the ADVISe cluster randomized controlled implementation trial. Addict Sci Clin Pract. 2015 Nov 19;10:26. doi: 10.1186/s13722-015-0047-0. PMID 26585638